CLINICAL TRIAL: NCT02379078
Title: Impact of an Interprofessional Shared Decision-making and Goal-setting Decision Aid for Patients With Diabetes - A Pilot Cluster Randomized Controlled Trial
Brief Title: Impact of an Interprofessional Shared Decision-making and Goal-setting Decision Aid for Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-014
Record Dates: First submitted 2015-02-11; First posted 2015-03-04 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
Keywords: Shared decision-making; Priority setting; Patient decision aid; Interprofessional care; Diabetes mellitus; Patient education; Medical informatics; Toolkit development; Study protocol; User-centred design; Qualitative methods
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shared decision-making aid (Experimental): At study start (step 1: provider-directed intervention phase): Online shared decision-making aid, 1-page provider enabler, provider training video made available to health care providers
  At 6 months (step 2: provider- and patient-directed phase): Online shared decision-making aid, 1-page patient enabler, patient training video also made available to patients (in addition to health care providers)
  Interventions: Other: Shared decision-making aid
- Generic hard-copy diabetes resources (Placebo Comparator): At study start (step 1: Provider-directed intervention phase): A hard copy of the executive summary of the CDA CPG and postcard outlining online resources made available to health care providers
  At 6 months (step 2: provider- and patient-directed phase): A CDA patient education pamphlet regarding diabetes self-management also made available to patients
  In addition, provider- and patient-directed guideline dissemination tools (not incorporating SDM) will also be publicly accessible from the CDA website.
  Interventions: Other: Generic hard copy diabetes resources; Other: Generic online diabetes resources

INTERVENTIONS:
Other: Shared decision-making aid — The IP-SDM toolkit consists of an online shared decision-making aid, 1-page provider enabler, a provider training video,1-page patient enabler, and a patient training video.
  Arms: Shared decision-making aid
Other: Generic hard copy diabetes resources — A hard copy of the executive summary of the CDA CPG and postcard outlining online resources, CDA patient education pamphlet
  Arms: Generic hard-copy diabetes resources
Other: Generic online diabetes resources — Provider- and patient-directed guideline dissemination tools (not incorporating SDM) publicly accessible from the CDA website
  Arms: Generic hard-copy diabetes resources

SUMMARY:
Diabetes care is complicated for people with diabetes as well as for health care providers: they have to watch their diet, exercise, take medications, checking blood sugars and blood pressure, get tests and see multiple doctors. On top of that, many with diabetes have other health problems, such as high blood pressure or arthritis, that make care even more complicated. Guidelines for improving the care of people with diabetes try to help by summarizing the best practices for care, but because diabetes care is so complicated, it is hard for them to be put into practice. One solution to this is a tool that can help people with diabetes set health care goals that are important to them, and participate actively in decisions about their own health care, together with health care providers. This tool would have an information booklet for patients with facts that can help them make a decision, a worksheet to help spell out what their goals are and how they want to get there, and a cheat-sheet for health care providers that gives them tips on how to do this. The purpose of this project is to find out if a tool like this would be helpful, how to make it more helpful and usable, and what the best way would be to make sure that people use it.

An interprofessional (IP) shared decision-making (SDM) and goal-setting tool kit, including a 1-page provider enabler, a point-of-care worksheet and a patient workbook, can be implemented successfully in clinical practice and will reduce decisional conflict and diabetes distress and improve chronic care delivery and quality of life in patients with type 1 or type 2 diabetes and 2 other comorbid chronic diseases. The investigators hypothesize that patients in the intervention arm of the study will have reduced decisional conflict and diabetes distress, and improved decision-making satisfaction, chronic care delivery and quality of life.

DETAILED DESCRIPTION:
Significance:

Diabetes is prevalent and results in major morbidity. Care of the patient with diabetes is complex and often occurs in the context of other chronic illness; this multimorbidity negatively impacts morbidity and mortality. The Canadian Diabetes Association (CDA) Clinical Practice Guidelines (CPG) are a rigorously developed knowledge tool that comprehensively address all aspects of diabetes care, conforming to AGREE II standards for guideline development. However, guideline adherence in the patient with multimorbidity is challenging both for the provider and the patient, who are overwhelmed by numerous, often conflicting recommendations. An individualized approach to the multimorbid diabetic patient using shared decision-making (SDM) and goal setting may overcome challenges to guideline adherence; however these strategies have not been taken up extensively in clinical practice. Barriers to uptake can be overcome by incorporating SDM into the context of interprofessional care: in diabetes care, role expansion, active participation by more than one discipline and adding additional team members have been demonstrated to improve clinical outcomes. While SDM and decision aids have typically focused on one issue, the precedent and potential exists for their use in the translation of the CDA CPG into practice through the prioritization of complex guideline recommendations. Given the growing prevalence of diabetes and multimorbidity in Canada, effectively bridging the knowledge to practice gap in this area has the potential to significantly improve patient-important outcomes, health care delivery and system sustainability.

Objectives:

1. To enhance the implementation of a complex guidelines document (CDA 2013 CPG) by assisting in prioritizing care for patients with diabetes and multiple other comorbidities through the use of a diabetes-focused SDM intervention;
2. To systematically develop, test and pilot a SDM and goal-setting intervention following the United Kingdom Medical Research Council and Knowledge to Action Frameworks;
3. To build a team consisting of members of the research community, patients, health care providers, CDA, and Local Health Integration Networks of the Ministry of Health and Long-Term Care, in order to increase the relevance of research conducted and enable dissemination of these research results into practice.

Hypothesis An interprofessional SDM and goal-setting tool kit, including a 1-page provider enabler, a point-of-care worksheet and a patient workbook, can be implemented successfully in clinical practice and will reduce decisional conflict and diabetes distress and improve chronic care delivery and quality of life in patients with type 1 or type 2 diabetes and 2 other comorbid chronic diseases.

Research Plan Development, testing and refinement: An evidence-based multi-component SDM intervention will be developed, framed by the Interprofessional SDM Model and based on user input from individual interviews regarding feasibility, acceptability and mediators of use. Usability testing will be done using cognitive task analysis to assess paths users take to accomplish tasks, errors made, when and where they encountered confusion or frustration, degree of satisfaction and quality of decision support. Based on feedback received, the tool will be refined through several iterative cycles of feedback and redesign.

Pilot trial: The tool kit will be piloted in a two-step parallel clustered randomized controlled trial (RCT) whose primary purpose is to assess intervention fidelity and to test the feasibility of conducting a larger RCT. The first step will be a provider-directed phase; the second step (which will occur 6 months later) will be a provider- and patient-directed phase. A secondary purpose of this study is to estimate the impact of the decision aid on decisional conflict; secondary outcomes include diabetes distress, chronic illness care and quality of life, assessed by patient-completed questionnaires of validated scales at baseline, 6 and 12 months. Analysis will be done by intention to treat. Multilevel hierarchical regression models will be used to account for the clustered nature of the data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Type 1 or Type 2 diabetes and
* have 2 or more other chronic comorbidities

Exclusion Criteria:

* do not speak English
* have documented cognitive deficits
* unable to give informed consent
* have limited life expectancy (<1 year)
* not available for follow-up
* seen primarily by a resident physician
* are pregnant or considering conception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Yu, MD FRCPC, Principal Investigator — St. Michael's Hospital (Unity Health Toronto)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu CH, Ivers NM, Stacey D, Rezmovitz J, Telner D, Thorpe K, Hall S, Settino M, Kaplan DM, Coons M, Sodhi S, Sale J, Straus SE. Impact of an interprofessional shared decision-making and goal-setting decision aid for patients with diabetes on decisional conflict--study protocol for a randomized controlled trial. Trials. 2015 Jun 27;16:286. doi: 10.1186/s13063-015-0797-8. PMID 26116444
- [Background] Yu CH, Stacey D, Sale J, Hall S, Kaplan DM, Ivers N, Rezmovitz J, Leung FH, Shah BR, Straus SE. Designing and evaluating an interprofessional shared decision-making and goal-setting decision aid for patients with diabetes in clinical care--systematic decision aid development and study protocol. Implement Sci. 2014 Jan 22;9:16. doi: 10.1186/1748-5908-9-16. PMID 24450385
- [Derived] Yu CH, Medleg F, Choi D, Spagnuolo CM, Pinnaduwage L, Straus SE, Cantarutti P, Chu K, Frydrych P, Hoang-Kim A, Ivers N, Kaplan D, Leung FH, Maxted J, Rezmovitz J, Sale J, Sodhi S, Stacey D, Telner D. Integrating shared decision-making into primary care: lessons learned from a multi-centre feasibility randomized controlled trial. BMC Med Inform Decis Mak. 2021 Nov 22;21(1):323. doi: 10.1186/s12911-021-01673-w. PMID 34809626
- [Derived] Yu CH, McCann M, Sale J. "In my age, we didn't have the computers": Using a complexity lens to understand uptake of diabetes eHealth innovations into primary care-A qualitative study. PLoS One. 2021 Jul 7;16(7):e0254157. doi: 10.1371/journal.pone.0254157. eCollection 2021. PMID 34234368
- [Derived] Yu C, Choi D, Bruno BA, Thorpe KE, Straus SE, Cantarutti P, Chu K, Frydrych P, Hoang-Kim A, Ivers N, Kaplan D, Leung FH, Maxted J, Rezmovitz J, Sale J, Sodhi-Helou S, Stacey D, Telner D. Impact of MyDiabetesPlan, a Web-Based Patient Decision Aid on Decisional Conflict, Diabetes Distress, Quality of Life, and Chronic Illness Care in Patients With Diabetes: Cluster Randomized Controlled Trial. J Med Internet Res. 2020 Sep 30;22(9):e16984. doi: 10.2196/16984. PMID 32996893
- [Derived] Yu CH, Ke C, Jovicic A, Hall S, Straus SE; IP-SDM Team;. Beyond pros and cons - developing a patient decision aid to cultivate dialog to build relationships: insights from a qualitative study and decision aid development. BMC Med Inform Decis Mak. 2019 Sep 18;19(1):186. doi: 10.1186/s12911-019-0898-5. PMID 31533828

RESULTS

PARTICIPANT FLOW:
Groups:
- Shared Decision-making Aid: At study start (step 1: provider-directed intervention phase): Online shared decision-making aid, 1-page provider enabler, provider training video made available to health care providers
  At 6 months (step 2: provider- and patient-directed phase): Online shared decision-making aid, 1-page patient enabler, patient training video also made available to patients (in addition to health care providers)
  Shared decision-making aid: The interprofessional (IP)-SDM toolkit consists of an online shared decision-making aid, 1-page provider enabler, a provider training video,1-page patient enabler, and a patient training video.
  Generic online diabetes resources: Provider- and patient-directed guideline dissemination tools (not incorporating SDM) publicly accessible from the Canadian Diabetes Association website
- Generic Hard-copy Diabetes Resources: At study start (step 1: Provider-directed intervention phase): A hard copy of the executive summary of the Canadian Diabetes Association (CDA) Clinical Practice Guidelines (CPG) and postcard outlining online resources made available to health care providers
  At 6 months (step 2: provider- and patient-directed phase): A CDA patient education pamphlet regarding diabetes self-management also made available to patients
  In addition, provider- and patient-directed guideline dissemination tools (not incorporating SDM) will also be publicly accessible from the CDA website.
  Generic hard copy diabetes resources: A hard copy of the executive summary of the CDA CPG and postcard outlining online resources, CDA patient education pamphlet
  Generic online diabetes resources: Provider- and patient-directed guideline dissemination tools (not incorporating SDM) publicly accessible from the CDA website
Period: Overall Study
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
Started | 111 | 114
Completed | 72 | 79
Not Completed | 39 | 35
Not completed — Lost to Follow-up | 33 | 30
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Shared Decision-making Aid: At study start (step 1: provider-directed intervention phase): Online shared decision-making aid, 1-page provider enabler, provider training video made available to health care providers
  At 6 months (step 2: provider- and patient-directed phase): Online shared decision-making aid, 1-page patient enabler, patient training video also made available to patients (in addition to health care providers)
  Shared decision-making aid: The IP-SDM toolkit consists of an online shared decision-making aid, 1-page provider enabler, a provider training video,1-page patient enabler, and a patient training video.
  Generic online diabetes resources: Provider- and patient-directed guideline dissemination tools (not incorporating SDM) publicly accessible from the CDA website
- Generic Hard-copy Diabetes Resources: At study start (step 1: Provider-directed intervention phase): A hard copy of the executive summary of the CDA CPG and postcard outlining online resources made available to health care providers
  At 6 months (step 2: provider- and patient-directed phase): A CDA patient education pamphlet regarding diabetes self-management also made available to patients
  In addition, provider- and patient-directed guideline dissemination tools (not incorporating SDM) will also be publicly accessible from the CDA website.
  Generic hard copy diabetes resources: A hard copy of the executive summary of the CDA CPG and postcard outlining online resources, CDA patient education pamphlet
  Generic online diabetes resources: Provider- and patient-directed guideline dissemination tools (not incorporating SDM) publicly accessible from the CDA website
- Total: Total of all reporting groups
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources | Total
Number analyzed (Participants) | 102 | 111 | 213
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-44 years | 2 | 7 | 9
  Age: 45-54 years | 11 | 9 | 20
  Age: 55-64 years | 20 | 28 | 48
  Age: 65-74 years | 47 | 38 | 85
  Age: 75-84 years | 16 | 24 | 40
  Age: 85+ years | 4 | 5 | 9
  Age: Undisclosed | 2 | 0 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth: Male | 46 | 65 | 111
  Sex at Birth: Female | 56 | 46 | 102
  Sex at Birth: Undisclosed | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White/Caucasian | 62 | 75 | 137
  Ethnicity: Black/African | 5 | 8 | 13
  Ethnicity: Asian | 19 | 8 | 27
  Ethnicity: Aboriginal | 4 | 3 | 7
  Ethnicity: Latin American | 1 | 2 | 3
  Ethnicity: Other | 7 | 15 | 22
  Ethnicity: Undisclosed | 4 | 0 | 4
Language [Count of Participants; unit: Participants]
  English | 81 | 103 | 184
  Other | 19 | 8 | 27
  Undisclosed | 2 | 0 | 2
Education [Count of Participants; unit: Participants]
  Bachelor | 23 | 17 | 40
  Below Bachelor | 3 | 5 | 8
  College | 30 | 26 | 56
  High School | 19 | 31 | 50
  Post-Grad | 13 | 12 | 25
  Below High School | 11 | 15 | 26
  Undisclosed | 3 | 5 | 8
Employment [Count of Participants; unit: Participants]
  Retired | 54 | 63 | 117
  Full time with employee health benefits | 22 | 15 | 37
  Full/part time without employee health benefits | 8 | 8 | 16
  Government assistance/disability | 3 | 6 | 9
  Unemployed | 2 | 5 | 7
  Stay at home parent, student or volunteer | 2 | 5 | 7
  Other | 7 | 4 | 11
  Prefer not to answer | 0 | 2 | 2
  Undisclosed | 4 | 3 | 7
Income [Count of Participants; unit: Participants]
  Less than $10k | 6 | 9 | 15
  $10-$19k | 6 | 18 | 24
  $20-$29k | 5 | 8 | 13
  $30-$39k | 7 | 13 | 20
  $40-$49k | 7 | 10 | 17
  $50-$59k | 5 | 8 | 13
  $60-$69k | 6 | 3 | 9
  $70-$79k | 6 | 6 | 12
  $80-$89k | 6 | 2 | 8
  $90-$99k | 6 | 8 | 14
  $100k-$149k | 8 | 7 | 15
  More than $150k | 11 | 11 | 22
  Undisclosed | 23 | 8 | 31
Living Arrangements [Count of Participants; unit: Participants]
  Alone | 26 | 30 | 56
  With family members | 28 | 24 | 52
  With partner/spouse | 38 | 46 | 84
  With roommates | 3 | 2 | 5
  Other | 6 | 8 | 14
  Undisclosed | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict in Patients With Diabetes
Description: Decisional conflict was chosen to allow us to assess the impact of our decision aid on the quality of the decision-making process, an important first measure of the effectiveness of a decision aid and the shared decision making process. This outcome is assessed by the Decisional Conflict Scale (DCS), a well-validated, patient-completed measure. DCS consists of 16 items, with 5 subscales (informed, values clarity, support, uncertainty, and effective decision) and an overall summary score. IT is scored on a 5-item Likert scale ranging from '0- strongly agree' to '4- strongly disagree'. It's minimum total score is 0 and it's maximum total score is 100. The higher the score, the worse the outcome. The lower the score, the better the outcome.
Time Frame: This outcome is measured at 0, 6 and 12 months.
Population: Patients with diabetes and 2 or more comorbidities.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
Number analyzed (Participants) | 102 | 111
score on a scale
  Baseline | 25.53 (14.73) | 23.56 (15.00)
  6 months | 21.97 (14.87) | 21.10 (12.79)
  12 months | 17.35 (11.21) | 19.58 (9.11)
Statistical Analysis 1: Comparison: Shared Decision-making Aid vs Generic Hard-copy Diabetes Resources; Test type: Superiority; p = 0.0246, Mixed Models Analysis

2. Secondary Outcome: Patient With Diabetes' Assessment of Their Chronic Illness Care
Description: This outcome was selected because it is a direct measure of knowledge use by patients that will allow us to better understand mediating variables of knowledge use such as patient activation, goal-setting, problem-solving, and decision support.
  This outcome is assessed by the Patient Assessment of Care for Chronic Conditions (PACIC), a well-validated patient-completed questionnaire. PACIC includes 20 items, scored on a 5 point Likert scale ranging from '1 - None of the time' to '5 - Always'. PACIC consists of 5 sub-scales (patient activation, delivery system design, goal setting, problem solving, and follow-up/coordination) and an overall summary score. The minimum total score is 0 and the maximum total score is 50. A higher score indicates a better outcome.
Time Frame: This outcome is measured at 0, 6 and 12 months.
Population: Patients with diabetes and 2 or more comorbidities.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
Number analyzed (Participants) | 111 | 102
score on a scale
  Baseline | 2.82 (1.10) | 3.16 (0.95)
  6 months | 3.16 (1.10) | 3.41 (1.05)
  12 months | 3.68 (0.99) | 3.22 (1.08)
Statistical Analysis 1: Comparison: Shared Decision-making Aid vs Generic Hard-copy Diabetes Resources; Test type: Superiority; p < 0.0001, Mixed Models Analysis

3. Secondary Outcome: Diabetes Distress in Patients With Diabetes
Description: This outcome was selected because it is a direct measure of knowledge use by patients that will allow us to better understand mediating variables of knowledge use such as patient activation, goal-setting, problem-solving, and decision support.
  This outcome is assessed by the Diabetes Distress Scale (DDS), a well-validated, patient-completed questionnaire. The DDS is a 17-item scale with 4 subscales (emotional burden, regimen distress, interpersonal distress and physician distress) with an overall summary score. It is scored on a 6-point Likert scale, ranging from '1 - no problem' to '6 - serious problem'. It's minimum total score is 0 and it's maximum total score is 6. The higher the score, the worse the outcome. The lower the score, the better the outcome.
Time Frame: This outcome is measured at 0, 6 and 12 months.
Population: Patients with diabetes and 2 or more comorbidities.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
Number analyzed (Participants) | 102 | 111
score on a scale
  Baseline | 2.08 (1.02) | 1.93 (0.83)
  6 months | 1.92 (1.09) | 1.88 (0.78)
  12 months | 1.86 (0.87) | 1.90 (0.75)
Statistical Analysis 1: Comparison: Shared Decision-making Aid vs Generic Hard-copy Diabetes Resources; Test type: Superiority; p = 0.12, Mixed Models Analysis

4. Secondary Outcome: Health-related Quality of Life in Patients With Diabetes
Description: Quality of life was selected to inform future sample size calculations, as more holistic and patient-centred measure of knowledge use that uniquely acknowledges patient prioritization of health care goals.
  This outcome is assessed by the Short Form 12 (SF-12), a well-validated, patient-completed questionnaire. The SF-12 consists of 12 items (minimum score is 0 and maximum score is 100; the higher the score, the better the quality of life.)
Time Frame: This outcome is measured at 0, 6 and 12 months.
Population: Patients with diabetes and 2 or more comorbidities.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
Number analyzed (Participants) | 102 | 111
score on a scale
  Baseline | 87.35 (14.25) | 89.69 (12.48)
  6 months | 88.88 (13.56) | 87.77 (12.87)
  12 months | 87.94 (12.87) | 86.99 (10.69)
Statistical Analysis 1: Comparison: Shared Decision-making Aid vs Generic Hard-copy Diabetes Resources; Test type: Superiority; p = 0.468, Mixed Models Analysis

5. Secondary Outcome: Intention to Engage in Shared Decision-making in Health Care Providers
Description: This outcome is assessed by the Continuing Professional Development (CPD) Reaction Questionnaire, a theory-based instrument to assess the impact of continuing professional development on clinical behavioral intentions. This outcome was selected to assess provider's intention to engage in shared decision-making, as a potential facilitator or barrier to shared decision-making. The CPD Reaction Questionnaire consists of 12 items with 5 subscales (intention, social influence, beliefs about capabilities, moral norm, and beliefs about consequences) and is scored on a 7-point Likert scale. It's minimum score is 1 and it's maximum score is 7. The higher the score, the better the outcome.
Time Frame: This outcome is measured at 0, 6 and 12 months.
Population: Clinicians
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
Number analyzed (Participants) | 29 | 24
score on a scale
  Baseline | 6.0 (0.7) | 6.0 (1.1)
  6 months | 6.0 (1.8) | 6.5 (0.6)
  12 months | 5.7 (1.4) | 6.0 (1.2)
Statistical Analysis 1: Comparison: Shared Decision-making Aid vs Generic Hard-copy Diabetes Resources; Test type: Superiority; p = 0.60, ANOVA

ADVERSE EVENTS:
Time Frame: Any adverse events monitored was collected over the length of the trial period of 12 months.
Description: The intervention, MyDiabetesPlan, is non-invasive web-based health tool aimed at facilitating conversations around diabetes management for patients and their health care providers. The intervention in this study is of low risk and participants in our study are not at risk for any serious adverse events or all-cause mortality.
Arm/Group | Shared Decision-making Aid | Generic Hard-copy Diabetes Resources
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/111
Other Adverse Events (participants affected / at risk) | 0/102 | 0/111

LIMITATIONS AND CAVEATS:
* Lack of blinding of participants (patients and clinicians) due to nature of the intervention
* Potential response bias (online and hard-copy survey)
* Attrition rate 29%
* Less than anticipated MyDiabetesPlan use
* Lack of clinical outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02379078/Prot_SAP_000.pdf